CLINICAL TRIAL: NCT06667986
Title: AI Rivals Traditional Bite Wing Radiography in Detecting Proximal Secondary Caries in A Group of Egyptian Patients at Cairo University, Faculty OF Dentistry Hospital (Diagnostic Accuracy Study)
Brief Title: Artificial Intellegence Rivals Digital Bitewing in Detect Secondary Caries
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Tallah Mohamed Mansour, general Practitioner at Health Administration, Faculty of Pharmacy, Cairo University, Cairo University
Other Study IDs: AI in detect dental caries
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Caries,Dental
Keywords: Secondary caries, Artificial intelligence, Digital bitewing radiography, Diagnostic accuracy study.
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: artificial intelligence models (YOLO and Mask-RCNN) — machine learning model will used to detect secondary caries around restorations by comparing the results with digital bitewing radiography

SUMMARY:
This study uses digital bitewing radiography as a standard for diagnosing proximal secondary caries. Patients will undergo imaging with a parallel technique and fixed settings to ensure high-quality, consistent images. Radiographs are interpreted by experienced dental professionals to maintain diagnostic accuracy. Machine learning models YOLO and Mask-RCNN will analyze these images in three phases: pre-analytical, analytical, and post-analytical. A dataset of 322 labeled images, annotated by experts, is used to train these models. Data augmentation methods enhance model performance, and accuracy is assessed against radiographic results to confirm reliability.

DETAILED DESCRIPTION:
Dental caries are chronic diseases that results in the destruction of the hard tooth tissues. It is a multifactorial condition that often goes undiagnosed, especially when it is hidden or in its initial stages. Detecting non-cavitated lesions is crucial for their early management. The standard visual-tactile inspection often fails to identify early lesions on hard-to-reach surfaces, such as proximal areas and beneath restorations. Detecting proximal caries early is crucial for implementing effective treatments and achieving optimal outcomes. A common supplementary method for detecting early lesions on proximal surfaces and assessing their extent is bitewing radiography. The routine diagnostic approach combines clinical examination with radiographic evaluation. To increase the detection rate of proximal secondary caries, experts recommend integrating visual and clinical examinations with bitewing radiography. Intraoral bitewing radiographs can be captured using either film or digital sensors, with preference for digital systems due to their benefits of reduced patient exposure, time savings, image enhancement, and ease of image storage, retrieval, and transmission. Although more sensitive for detecting early lesions than visual-tactile assessments, bitewing evaluations comes with significant variance between examiners and a considerable proportion of false-positive or false-negative detections. Recent literature has explored the use of artificial intelligence (AI), a field of computer science focused on developing machines capable of mimicking human cognitive abilities, as a diagnostic tool for detecting caries lesions using dental (digital radiographic) images. As AI technology advances, an increasing number of studies have examined the diagnostic performance of AI-based models, emphasizing the importance of creating reliable tools like AI to enhance the diagnostic process. Numerous studies have assessed the performance of AI models on diverse types of dental radiographs, with a significant focus on bitewing radiographs (BWR). AI has been used for various applications in oral and dental health, including the detection of dental caries, endodontic treatment and diagnosis, periodontal issues, and the detection of oral lesion pathology. A reference dataset of caries diagnoses from bitewing radiographs by different examiners created this benchmark which serves as a crucial tool for comparing the diagnostic performance of AI models against human examiners, emphasizing the potential improvements in accuracy and reliability that AI can bring to dental diagnostics.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients Aged 22-60 Patient
2. Males or females.
3. Patients have proximal restorations.
4. Co-operative patients who show interest in participating in the study.

Exclusion Criteria:

1. Patients with orthodontic appliances, or bridge work that might interfere with evaluation
2. Patients with no caries.
3. Systematic disease that may affect participation.
4. Patients not willing to be part of the study or ones who refuse to sign the informed consent.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients attending the Conservative Department at Cairo University Dental Clinic who present with proximal restorations, show no signs or symptoms, demonstrate cooperation, and express interest in participating in the study will be considered eligible. Patients with orthodontic appliances or bridgework that could impact the quality of radiographic imaging will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
two deep learning models, YOLO and Mask-RCNN, will be trained on this dataset to accurately detect and classify images showing signs of secondary caries | baseline
  models will detect the presence or absence of secondary caries around restorations

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Heba Hamza, professor, Study Director — Professor of Conservative Dentistry Department, Faculty of Dentistry, Cairo University; Dr. Rawda Hisham A. ElAziz, lecturer, Study Director — Lecturer of Conservative Dentistry Department, Faculty of Dentistry, Cairo University; Dr. Asmaa Ahmed Elsayed Osman, lecturer, Study Director — Lecturer of Information Technology, Faculty of Computers and Artificial Intelligence, Cairo University

REFERENCES:
- [Result] Chaves ET, Vinayahalingam S, van Nistelrooij N, Xi T, Romero VHD, Flugge T, Saker H, Kim A, Lima GDS, Loomans B, Huysmans MC, Mendes FM, Cenci MS. Detection of caries around restorations on bitewings using deep learning. J Dent. 2024 Apr;143:104886. doi: 10.1016/j.jdent.2024.104886. Epub 2024 Feb 9. PMID 38342368
- [Result] Mohammad-Rahimi H, Motamedian SR, Rohban MH, Krois J, Uribe SE, Mahmoudinia E, Rokhshad R, Nadimi M, Schwendicke F. Deep learning for caries detection: A systematic review. J Dent. 2022 Jul;122:104115. doi: 10.1016/j.jdent.2022.104115. Epub 2022 Mar 30. PMID 35367318
- [Result] Mertens S, Krois J, Cantu AG, Arsiwala LT, Schwendicke F. Artificial intelligence for caries detection: Randomized trial. J Dent. 2021 Dec;115:103849. doi: 10.1016/j.jdent.2021.103849. Epub 2021 Oct 14. PMID 34656656
- [Result] Chen X, Guo J, Ye J, Zhang M, Liang Y. Detection of Proximal Caries Lesions on Bitewing Radiographs Using Deep Learning Method. Caries Res. 2022;56(5-6):455-463. doi: 10.1159/000527418. Epub 2022 Oct 10. PMID 36215971